CLINICAL TRIAL: NCT01764529
Title: Modifiers of Disease Severity and Progression in Cerebral Cavernous Malformations
Brief Title: Modifiers of Disease Severity in Cerebral Cavernous Malformations
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: University of New Mexico (Other); University of Chicago (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Boston Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Barrow Neurological Institute (Other); Alliance to Cure Cavernous Malformation (Unknown)
Responsible Party: Sponsor
Other Study IDs: BVMC 6201; U54NS065705-15 (NIH)
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Cavernous Angioma, Familial; Cerebral Cavernous Malformations; Cerebral Cavernous Hemangioma
MeSH Terms: conditions — Hemangioma, Cavernous, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Biospecimen Retention: Samples With DNA — We will collect stool specimens in newly recruited familial CCM cases. We collect and store saliva as well as whole blood for DNA, RNA, and plasma or serum samples. Brain cavernous malformation tissue will be collected and banked as available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The BVMC FCCM cohort: Aim 1: To investigate the relationship between lesion burden and outcomes in familial CCM.
  Aim 2: To investigate the role of the gut microbiome in familial CCM disease severity.
  Aim 3: To establish blood markers predictive of disease severity and progression for medical treatment of CCM.

SUMMARY:
Cerebral cavernous malformations (CCMs) are clusters of abnormal blood vessels in the brain and spine. CCMs can bleed and cause strokes, seizures, and headaches. CCMs are often caused by an inherited gene mutation (alteration) in one of three CCM genes (CCM1, CCM2, or CCM3). There is a wide range of disease severity even among family members with this disease, though the natural history has not been clearly described for this particular population.

This study will continue to enroll and follow participants with familial CCM to identify factors that influence CCM disease severity and progression, focusing on barriers to clinical trial preparedness. Our long-term goal is to identify measurable outcomes and robust biomarkers that will help select high-risk patients and help monitor drug response in future clinical trials.

The specific goals of this study are to:

* Identify factors that influence lesion progression to symptomatic hemorrhage and other outcomes, including quality of life;
* Investigate the role of the gut microbiome and lesion burden in CCM disease, and
* Identify blood biomarkers predictive of CCM disease severity and progression for clinical trials.

DETAILED DESCRIPTION:
This study is one of three projects participating in the Brain Vascular Malformation Consortium (BVMC) funded by the Office of Rare Diseases Research, which is part of the National Center for Advancing Translational Sciences (NCATS), and the National Institute of Neurological Disorders and Stroke (NINDS).

The CCM project is a cross-sectional and longitudinal study of familial CCM patients. The study is currently in the third 5-year cycle. During the first 5 year cycle (BVMC1), the CCM project was focused on recruiting CCM1 cases with the common Hispanic mutation (CHM). In the second 5-year cycle (BVMC2), we expanded recruitment to include not only CCM1-CHM cases, but also other CCM familial patients and mutation carriers. In the third 5-year cycle (BVMC3), we will continue to recruit familial CCM cases and expand to additional recruitment sites.

We collect clinical, genetic, imaging, treatment, and outcome data in participants, and follow enrolled participants over time to understand the natural history of this disease.

For new study participants, you will be asked to:

* Give permission for study staff to access your medical records to collect clinical information and to obtain copies of MRI scans and reports.
* Fill out a questionnaire about your quality of life, family history, and medical/surgical history.
* Give a blood and/or saliva sample, and stool sample.
* Give permission to store and use your CCM resected tissue for research (if undergoing surgery).
* Participate in annual follow-ups to update medical, surgical, and neurological information.

Eligible cases include those with a known genetic mutation in one of the three CCM genes or those that meet 2 of 3 following clinical criteria:

1. Clinical diagnosis of CCM,
2. Multi-focal lesions on MRI, and/or
3. Family history of CCMs.

Exclusion Criteria:

1. Patients who cannot or are unwilling to sign informed consent and for whom no appropriate surrogate is available.
2. Prisoners and homeless individuals because of the inability to contact the subject and collect follow-up data using standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Individual has a CCM mutation confirmed through DNA testing, or
* Individual meets 2 or more of the following clinical criteria:

  1. Clinical diagnosis of CCM
  2. Multi-focal CCMs on MRI
  3. Family history of CCM

Exclusion Criteria:

1. Individuals who are incarcerated
2. Individuals who are homeless
3. Unable or unwilling to sign the informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals who carry the diagnosis of familial cerebral cavernous malformation (CCM), both symptomatic and asymptomatic.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-04-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Total CCM lesion number per patient | Baseline
  The number of lesions (or cavernous angiomas) located in the brain will be counted by a neuroradiologist and by an automated algorithm developed as part of this project.
Rate of symptomatic hemorrhage | Baseline and annual assessment
  Symptomatic hemorrhage is defined as diagnostic evidence of new lesional bleeding or hemorrhagic growth, in association with directly attributable symptoms. Rate of symptomatic hemorrhage and the factors that influence hemorrhage rates will be assessed.

SECONDARY OUTCOMES:
Change in lesion number | Baseline, Follow up MRI
  The number of lesions (or cavernous angiomas) counted on the baseline MRI will be compared to the number of lesions observed in follow up MRIs.
Modified Rankin score | Baseline and annual assessment
  The modified Rankin score will be assessed at baseline and at approximately one year intervals while remaining in study

OTHER OUTCOMES:
Patient-Reported Quality of Life (QoL) (NIH PROMIS-29) | Baseline and annual assessment
  Standardized patient reported outcome measurement tools to assess pain, fatigue, physical function, emotional distress, and social participation.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Kim, PhD, Principal Investigator — University of California, San Francisco; Issam Awad, MD, Principal Investigator — University of Chicago
Locations (7):
- United States (7):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California, San Francisco, San Francisco, California
  - University of Chicago, Medicine and Biological Sciences, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Cincinnati Children's Hospital, Division of Pediatric Neurosurgery, Cerebrovascular Program, Cincinnati, Ohio
  - Alliance to Cure Cavernous Malformation, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Available data will be released to the Rare Diseases Clinical Research Network repository and will become available to the scientific community one year after publication of planned analyses, or after a period of 5 years from the date when the data were collected, whichever comes first

REFERENCES:
- [Background] Akers AL, Ball KL, Clancy M, Comi AM, Faughnan ME, Gopal-Srivastava R, Jacobs TP, Kim H, Krischer J, Marchuk DA, McCulloch CE, Morrison L, Moses M, Moy CS, Pawlikowska L, Young WL. Brain Vascular Malformation Consortium: Overview, Progress and Future Directions. J Rare Disord. 2013 Apr 1;1(1):5. PMID 25221778
- [Background] Flemming KD, Smith E, Marchuk D, Derry WB. Familial Cerebral Cavernous Malformations. 2003 Feb 24 [updated 2023 Jul 27]. In: Adam MP, Bick S, Mirzaa GM, Pagon RA, Wallace SE, Amemiya A, editors. GeneReviews(R) [Internet]. Seattle (WA): University of Washington, Seattle; 1993-2026. Available from http://www.ncbi.nlm.nih.gov/books/NBK1293/ PMID 20301470
- [Background] Choquet H, Pawlikowska L, Lawton MT, Kim H. Genetics of cerebral cavernous malformations: current status and future prospects. J Neurosurg Sci. 2015 Sep;59(3):211-20. Epub 2015 Apr 22. PMID 25900426
- [Background] Zafar A, Quadri SA, Farooqui M, Ikram A, Robinson M, Hart BL, Mabray MC, Vigil C, Tang AT, Kahn ML, Yonas H, Lawton MT, Kim H, Morrison L. Familial Cerebral Cavernous Malformations. Stroke. 2019 May;50(5):1294-1301. doi: 10.1161/STROKEAHA.118.022314. No abstract available. PMID 30909834
- [Background] Hart BL, Mabray MC, Morrison L, Whitehead KJ, Kim H. Systemic and CNS manifestations of inherited cerebrovascular malformations. Clin Imaging. 2021 Jul;75:55-66. doi: 10.1016/j.clinimag.2021.01.020. Epub 2021 Jan 20. PMID 33493737
- [Result] Choquet H, Pawlikowska L, Nelson J, McCulloch CE, Akers A, Baca B, Khan Y, Hart B, Morrison L, Kim H; Brain Vascular Malformation Consortium (BVMC) Study. Polymorphisms in inflammatory and immune response genes associated with cerebral cavernous malformation type 1 severity. Cerebrovasc Dis. 2014;38(6):433-40. doi: 10.1159/000369200. Epub 2014 Dec 3. PMID 25472749
- [Result] Choquet H, Nelson J, Pawlikowska L, McCulloch CE, Akers A, Baca B, Khan Y, Hart B, Morrison L, Kim H. Association of cardiovascular risk factors with disease severity in cerebral cavernous malformation type 1 subjects with the common Hispanic mutation. Cerebrovasc Dis. 2014;37(1):57-63. doi: 10.1159/000356839. Epub 2013 Dec 21. PMID 24401931
- [Result] Golden M, Saeidi S, Liem B, Marchand E, Morrison L, Hart B. Sensitivity of patients with familial cerebral cavernous malformations to therapeutic radiation. J Med Imaging Radiat Oncol. 2015 Feb;59(1):134-6. doi: 10.1111/1754-9485.12269. Epub 2015 Jan 7. PMID 25565562
- [Result] Hart BL, Taheri S, Rosenberg GA, Morrison LA. Dynamic contrast-enhanced MRI evaluation of cerebral cavernous malformations. Transl Stroke Res. 2013 Oct;4(5):500-6. doi: 10.1007/s12975-013-0285-y. Epub 2013 Sep 21. PMID 24323376
- [Result] Petersen TA, Morrison LA, Schrader RM, Hart BL. Familial versus sporadic cavernous malformations: differences in developmental venous anomaly association and lesion phenotype. AJNR Am J Neuroradiol. 2010 Feb;31(2):377-82. doi: 10.3174/ajnr.A1822. Epub 2009 Oct 15. PMID 19833796
- [Result] Choquet H, Trapani E, Goitre L, Trabalzini L, Akers A, Fontanella M, Hart BL, Morrison LA, Pawlikowska L, Kim H, Retta SF. Cytochrome P450 and matrix metalloproteinase genetic modifiers of disease severity in Cerebral Cavernous Malformation type 1. Free Radic Biol Med. 2016 Mar;92:100-109. doi: 10.1016/j.freeradbiomed.2016.01.008. Epub 2016 Jan 19. PMID 26795600
- [Result] Golden MJ, Morrison LA, Kim H, Hart BL. Increased number of white matter lesions in patients with familial cerebral cavernous malformations. AJNR Am J Neuroradiol. 2015 May;36(5):899-903. doi: 10.3174/ajnr.A4200. Epub 2015 Jan 2. PMID 25556204
- [Result] Zou X, Hart BL, Mabray M, Bartlett MR, Bian W, Nelson J, Morrison LA, McCulloch CE, Hess CP, Lupo JM, Kim H. Automated algorithm for counting microbleeds in patients with familial cerebral cavernous malformations. Neuroradiology. 2017 Jul;59(7):685-690. doi: 10.1007/s00234-017-1845-8. Epub 2017 May 22. PMID 28534135
- [Result] Strickland CD, Eberhardt SC, Bartlett MR, Nelson J, Kim H, Morrison LA, Hart BL. Familial Cerebral Cavernous Malformations Are Associated with Adrenal Calcifications on CT Scans: An Imaging Biomarker for a Hereditary Cerebrovascular Condition. Radiology. 2017 Aug;284(2):443-450. doi: 10.1148/radiol.2017161127. Epub 2017 Mar 20. PMID 28318403
- [Result] Akers A, Al-Shahi Salman R, A Awad I, Dahlem K, Flemming K, Hart B, Kim H, Jusue-Torres I, Kondziolka D, Lee C, Morrison L, Rigamonti D, Rebeiz T, Tournier-Lasserve E, Waggoner D, Whitehead K. Synopsis of Guidelines for the Clinical Management of Cerebral Cavernous Malformations: Consensus Recommendations Based on Systematic Literature Review by the Angioma Alliance Scientific Advisory Board Clinical Experts Panel. Neurosurgery. 2017 May 1;80(5):665-680. doi: 10.1093/neuros/nyx091. PMID 28387823
- [Result] Tang AT, Choi JP, Kotzin JJ, Yang Y, Hong CC, Hobson N, Girard R, Zeineddine HA, Lightle R, Moore T, Cao Y, Shenkar R, Chen M, Mericko P, Yang J, Li L, Tanes C, Kobuley D, Vosa U, Whitehead KJ, Li DY, Franke L, Hart B, Schwaninger M, Henao-Mejia J, Morrison L, Kim H, Awad IA, Zheng X, Kahn ML. Endothelial TLR4 and the microbiome drive cerebral cavernous malformations. Nature. 2017 May 18;545(7654):305-310. doi: 10.1038/nature22075. Epub 2017 May 10. PMID 28489816
- [Result] Morrison MA, Payabvash S, Chen Y, Avadiappan S, Shah M, Zou X, Hess CP, Lupo JM. A user-guided tool for semi-automated cerebral microbleed detection and volume segmentation: Evaluating vascular injury and data labelling for machine learning. Neuroimage Clin. 2018 Aug 4;20:498-505. doi: 10.1016/j.nicl.2018.08.002. eCollection 2018. PMID 30140608
- [Result] Mabray MC, Caprihan A, Nelson J, McCulloch CE, Zafar A, Kim H, Hart BL, Morrison L. Effect of Simvastatin on Permeability in Cerebral Cavernous Malformation Type 1 Patients: Results from a Pilot Small Randomized Controlled Clinical Trial. Transl Stroke Res. 2020 Jun;11(3):319-321. doi: 10.1007/s12975-019-00737-4. Epub 2019 Oct 23. No abstract available. PMID 31643041
- [Result] Tang AT, Sullivan KR, Hong CC, Goddard LM, Mahadevan A, Ren A, Pardo H, Peiper A, Griffin E, Tanes C, Mattei LM, Yang J, Li L, Mericko-Ishizuka P, Shen L, Hobson N, Girard R, Lightle R, Moore T, Shenkar R, Polster SP, Rodel CJ, Li N, Zhu Q, Whitehead KJ, Zheng X, Akers A, Morrison L, Kim H, Bittinger K, Lengner CJ, Schwaninger M, Velcich A, Augenlicht L, Abdelilah-Seyfried S, Min W, Marchuk DA, Awad IA, Kahn ML. Distinct cellular roles for PDCD10 define a gut-brain axis in cerebral cavernous malformation. Sci Transl Med. 2019 Nov 27;11(520):eaaw3521. doi: 10.1126/scitranslmed.aaw3521. PMID 31776290
- [Result] Tandberg SR, Bocklage T, Bartlett MR, Morrison LA, Nelson J, Hart BL. Vertebral Intraosseous Vascular Malformations in a Familial Cerebral Cavernous Malformation Population: Prevalence, Histologic Features, and Associations With CNS Disease. AJR Am J Roentgenol. 2020 Feb;214(2):428-436. doi: 10.2214/AJR.19.21492. Epub 2019 Dec 11. PMID 31825263
- [Result] Manole AK, Forrester VJ, Zlotoff BJ, Hart BL, Morrison LA. Cutaneous findings of familial cerebral cavernous malformation syndrome due to the common Hispanic mutation. Am J Med Genet A. 2020 May;182(5):1066-1072. doi: 10.1002/ajmg.a.61519. Epub 2020 Feb 26. PMID 32100472
- [Result] Campbell R, Petranovich CL, Cheek S, Morrison L, Hart B. Subjective Cognitive Concerns and Attitudes toward Genetic Testing Are Associated with Depressive Symptoms and Quality of Life after Genetic Testing for the Cerebral Cavernous Malformation Common Hispanic Mutation (CCM1). J Behav Brain Sci. 2020 Feb;10(2):118-127. doi: 10.4236/jbbs.2020.102007. Epub 2020 Feb 25. PMID 32467778
- [Result] Mabray MC, Starcevich J, Hallstrom J, Robinson M, Bartlett M, Nelson J, Zafar A, Kim H, Morrison L, Hart BL. High Prevalence of Spinal Cord Cavernous Malformations in the Familial Cerebral Cavernous Malformations Type 1 Cohort. AJNR Am J Neuroradiol. 2020 Jun;41(6):1126-1130. doi: 10.3174/ajnr.A6584. Epub 2020 May 28. PMID 32467184
- [Result] Polster SP, Sharma A, Tanes C, Tang AT, Mericko P, Cao Y, Carrion-Penagos J, Girard R, Koskimaki J, Zhang D, Stadnik A, Romanos SG, Lyne SB, Shenkar R, Yan K, Lee C, Akers A, Morrison L, Robinson M, Zafar A, Bittinger K, Kim H, Gilbert JA, Kahn ML, Shen L, Awad IA. Permissive microbiome characterizes human subjects with a neurovascular disease cavernous angioma. Nat Commun. 2020 May 27;11(1):2659. doi: 10.1038/s41467-020-16436-w. PMID 32461638
- [Result] Weinsheimer S, Nelson J, Abla AA, Ko NU, Tsang C, Okoye O, Zabramski JM, Akers A, Zafar A, Mabray MC, Hart BL, Morrison L, McCulloch CE, Kim H; Brain Vascular Malformation Consortium Cerebral Cavernous Malformation Investigator Group *. Intracranial Hemorrhage Rate and Lesion Burden in Patients With Familial Cerebral Cavernous Malformation. J Am Heart Assoc. 2023 Feb 7;12(3):e027572. doi: 10.1161/JAHA.122.027572. Epub 2023 Jan 25. PMID 36695309
- [Result] Fox CK, Nelson J, McCulloch CE, Weinsheimer S, Pawlikowska L, Hart B, Mabray MC, Zafar A, Morrison L, Zabramski JM, Akers A, Kim H. Seizure Incidence Rates in Children and Adults With Familial Cerebral Cavernous Malformations. Neurology. 2021 Sep 20;97(12):e1210-e1216. doi: 10.1212/WNL.0000000000012569. PMID 34389651
- [Result] Choksi F, Weinsheimer S, Nelson J, Pawlikowska L, Fox CK, Zafar A, Mabray MC, Zabramski J, Akers A, Hart BL, Morrison L, McCulloch CE, Kim H. Assessing the association of common genetic variants in EPHB4 and RASA1 with phenotype severity in familial cerebral cavernous malformation. Mol Genet Genomic Med. 2021 Oct;9(10):e1794. doi: 10.1002/mgg3.1794. Epub 2021 Sep 7. PMID 34491620
- [Result] Wetzel-Strong SE, Weinsheimer S, Nelson J, Pawlikowska L, Clark D, Starr MD, Liu Y, Kim H, Faughnan ME, Nixon AB, Marchuk DA. Pilot investigation of circulating angiogenic and inflammatory biomarkers associated with vascular malformations. Orphanet J Rare Dis. 2021 Sep 3;16(1):372. doi: 10.1186/s13023-021-02009-7. PMID 34479577
- See also: Angioma Alliance is an organization by and for those affected by cavernous angiomas and their loved ones, health professionals, and researchers. — https://www.alliancetocure.org